CLINICAL TRIAL: NCT04213118
Title: An Open, Single Arm,Multicenter Clinical Trial of Anlotinib Combined With Transcatheter Arterial Chemoembolization for Adjuvant Therapy in Patients With High Risk of Recurrence After Resection of Advanced Hepatocellular Carcinoma
Brief Title: Anlotinib Combined With TACE in Hepatocellular Carcinoma Patients at High Risk of Post Surgery Recurrence
Acronym: ALTER-H-004
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLLSL-2019-185
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma; TACE; Anlotinib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Administration anlotinib and it should be continued until relapse of HCC or intolerable toxicity or patients withdrawal of consent.
  Interventions: Drug: Anlotinib Hydrochloride; Procedure: TACE

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib 12mg QD PO d1-14, 21 days per cycle.
Procedure: TACE — TACE first, followed by anlotinib within day4（+/-1days）

SUMMARY:
A single-arm, open-label clinical trial to assess the effects and safety of anlotinib hydrochloride combined with transcatheter arterial chemoembolization (TACE) in hepatocellular carcinoma(HCC) patients at high risk of post surgery recurrence.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most common malignant tumors in the world with high incidence and mortality. Recurrence of HCC is still a great challenge and threat to the patients after resection surgery. Anlotinib is a new, orally administered tyrosine kinase inhibitor that targets vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptors (PDGFR), and c-kit.

HCC patients who meet the eligibility criteria of this clinical trial will adopt postoperative TACE combined with anlotinib hydrochloride. At Day4 of TACE,anlotinib 12mg QD PO d1-14, 21 days per cycle until disease progresses or intolerant.

Primary Efficacy Endpoint: Disease free survival (DFS);Secondary Efficacy Endpoints: 1-year DFS Rate and Time to recurrence (TTR)(According to RECIST Version 1.1).Safety will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients participate in the study voluntarily and sign informed consent with good compliance.
* After hepatectomy, satisfy any of the following recurrence factors was assessed:≥5 cm and < 10 cm of tumor diameter; tumor number≥3; tumor microvascular invasion grade M1; portal vein carcinoma thrombus resection(Ⅰ、Ⅱ).
* Histological or cytological confirmation of hepatocellular carcinoma, or at least two imaging tests with hepatocellular carcinoma characteristics, or one imaging test with hepatocellular carcinoma characteristics and AFP > 400μg/L.
* TACE treatment (cTACE only) was completed within 1-2 months after hepatectomy.
* ≥ 18 and ≤ 75 years of age.
* ECOG performance status of 0-1.
* liver function child-Pugh class A or B (≤7 points).
* Except for hepatectomy, no previous tumor-related treatment was received, and the remaining liver was assessed to have good liver function.

Exclusion Criteria:

* Patients who have had or are currently complicated with other malignant tumors,or recurrent hepatocellular carcinoma (>10 mm)in baseline data or in TACE.
* Patients with absolute contraindications to TACE.
* Patients with HCV infection.
* Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed.
* Pregnant or lactating women.
* Patients with mental illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From randomization to recurrence of HCC or death (up to 1year)
  The period from resection surgery to recurrence of HCC

SECONDARY OUTCOMES:
1-year DFS Rate | From randomization to recurrence of HCC or death (up to 1year)
  One year ratio of DFS
Time to recurrence | From randomization to recurrence of HCC(up to 1year)
  The period from resection surgery to recurrence of HCC
Incidence of Treatment-Emergent Adverse Events Safety and Tolerability | Up to 30 day safety follow-up visit
  Any adverse effects occur during the use of anlotinib

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wu, PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (4):
- China (4):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Hanzhong Central Hospital, Hanzhong, Shaanxi
  - Tangdu Hospital of The Fourth Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

REFERENCES:
- [Derived] Wang Z, Zhang L, Zheng X, Zhang D, Yang X, Xu K, Tao J, Song X, Ma J, Wu Z. Adjuvant anlotinib plus TACE in hepatocellular carcinoma with postoperative high-risk recurrence: a single-arm, multi-center, phase II study. Clin Transl Oncol. 2026 Jan 3. doi: 10.1007/s12094-025-04160-0. Online ahead of print. PMID 41484570